CLINICAL TRIAL: NCT06523140
Title: Management of Chronic Obstructive Pulmonary Disease (COPD) Patients With BoraCare® Remote Monitoring Solution Including BVS3 Early Detection Score for COPD Exacerbations
Brief Title: Management of COPD Patients With BoraCare® Remote Monitoring Solution Including BVS3 Early Detection Score for COPD Exacerbations
Acronym: AUSTRAAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biosency (Industry)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-A02454-41
Record Dates: First submitted 2024-07-08; First posted 2024-07-26 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: COPD
Keywords: Remote monitoring; COPD; Prevention; Exacerbations; Patient quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Comparative, superior, randomised, multicentre, two-arm study (experimental group, control group, 1:1 ratio) in open-label, with a pilot phase
  Control group:
  Conventional follow-up: two consultations with the general practitioner and one consultation with the pulmonologist per year. The inclusion and follow-up visit at 12 months by a pulmonologist are consistent with the follow-up of COPD patients in current practice and the recommendations of SAH and SPLF.
  Experimental group:
  Patients will receive conventional clinical follow-up and at the same time benefit from the Bora care remote monitoring system. Patients are monitored daily remotely by Case Managers, who, when the BVS3-3 alarm is triggered on Bora Connect, call the patient to inform the patient about his symptoms, then notify the pulmonologist by transmitting the information from Bora Connect. The Case Manager re-evaluates the situation at 48h and 96h if necessary and forwards the information to the pulmonologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Conventional follow-up: two consultations with the general practitioner and one consultation with the pulmonologist per year. The inclusion and follow-up visit at 12 months by a pulmonologist are consistent with the follow-up of COPD patients in current practice and the recommendations of SAH and SPLF.
- Experimental group (Experimental): Patients will receive conventional clinical follow-up and at the same time benefit from the Bora care remote monitoring system. Patients are monitored daily remotely by Case Managers, who, when the BVS3-3 alarm is triggered on Bora Connect, call the patient to inform the patient about his symptoms, then notify the pulmonologist by transmitting the information from Bora Connect and the minutes of the phone call, who, according to conventional management, decides whether or not to hospitalize the patient, or to generate an unscheduled consultation in order to prescribe drug treatment, and/or to prescribe additional examinations, and/or to adapt the patient's oxygen therapy prescription. The Case Manager re-evaluates the situation at 48h and 96h if necessary and forwards the information to the pulmonologist.
  Interventions: Device: Boracare remote monitoring solution

INTERVENTIONS:
Device: Boracare remote monitoring solution — Bora Band wristband measuring vital signs at home, Bora Connect platform for caregiver visualization and BVS3 early detection of COPD exacerbations
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to demonstrate the superiority of remote monitoring with the Bora Care solution in patients with COPD and frequent exacerbations (experimental group) compared to conventional follow-up alone (control group) on the total number of hospital days per patient for respiratory deterioration over 12 months of follow-up.

The main question it aims to answer is: Does remote monitoring of COPD patients reduce the average annual length of hospitalization for exacerbations of COPD patients?

All participants will benefit a conventional clinical follow-up.

Participants in experimental group will also benefit from the Bora care remote monitoring system.

DETAILED DESCRIPTION:
Control group (control): conventional follow-up For the target population (frequent exacerbating COPD patients), the usual follow-up includes two consultations with the general practitioner and one consultation with the pulmonologist per year. The inclusion and follow-up visit at 12 months by a pulmonologist are consistent with the follow-up of COPD patients in current practice and the recommendations of HAS (National Authority for Health) and SPLF (French-Language Society of Pneumology).

Experimental group (conventional monitoring + remote monitoring):

The patients will be subject to conventional clinical follow-up and at the same time benefit from the Bora care remote monitoring system. The Bora care remote monitoring system includes a BoraBand wristband measuring vital signs at home, the Bora Connect platform for caregiver visualization of data and the BVS3 score for early detection of COPD exacerbations. Patients are monitored daily remotely by Case Managers (nurses trained in Bora Care solution), who, when the BVS3 > 3 alert is triggered on Bora Connect, call the patient to inform the patient about his symptoms, then alert the pulmonologist by transmitting the information from Bora Connect and the minutes of the phone call, who, according to conventional management, decides whether or not to hospitalize the patient, or to generate an unscheduled consultation in order to prescribe drug treatment, and/or to prescribe additional examinations, and/or to adapt the patient's oxygen therapy prescription.

The Case Manager re-evaluates the situation after 48 hours and 96 hours if necessary and forwards the information to the pulmonologist. The nature of the transmission of information (telephone or email) between the Case Manager and the pulmonologist in case of an alert is defined when the patient is included by the pulmonologist. If desired, remotely monitored patients will be able to access the Bora Connect interface provided for patients (restricted viewing of data).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age with COPD defined according to the recommendations of the SPLF, whose level of respiratory function in a stable state is known (measured less than 12 months), recruited in pulmonology
* Patient who has been hospitalized for COPD exacerbation in the previous 12 months
* Informed patient who has signed consent,
* Patient enrolled in a social security scheme (Art L1121-11 of the CSP)

Exclusion Criteria:

* Presence of a comorbidity considered unstable or very severe by the investigator.
* Patient with psychological frailties,
* Patient already included in another interventional trial,
* Patient who does not speak French and is unable to use the Bora Band tool and without access to a caregiver,
* Patient protected under guardianship or unable to give free and informed consent.
* Pregnant or nursing woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the superiority of remote monitoring with the Bora Care solution in patients with COPD and frequent exacerbations compared to conventional follow-up. | 1 year
  Number of hospital days for respiratory deterioration per patient over 12 months.

SECONDARY OUTCOMES:
Evaluate the effect of the device on the number of hospitalizations per patient. | 1 year
  Number of hospitalizations within 12 months of implementation of Bora Care remote monitoring.
Evaluate the effect of the device on the average length of stay. | 1 year
  Average length of stay in hospital within 12 months of the implementation of Bora Care.
Assess the overall quality of life of patients at baseline and at the end of the trial. (1) | 1 year
  Score from CAT (Chronic Obstructive Pulmonary Disease Assessment Test) questionnaire to assess the quality of life collected at Day 0, M6, M12.
Assess the overall quality of life of patients at baseline and at the end of the trial. (2) | 1 year
  Score from Short Form 36 (SF36) quality of life assessment questionnaire to assess the quality of life collected at Day 0, M6, M12.
Assess the overall quality of life of patients at baseline and at the end of the trial. (3) | 1 year
  Score from EXACT E-RS (Evaluating Respiratory Symptoms) symptom assessment questionnaire to assess the quality of life collected at Day 0, M6, M12.
Assess the conformity of use of the Bora Care device. | 3 years
  Number of hours spent wearing the Bora Connect bracelet normalized by the total number of hours spent in the remote monitoring session, information collected via the Bora Care tool.
Assess the impact of the device on the organisation of care. (1) | 3 years
  Number and nature of emergency, resuscitation, consultations and teleconsultations with the pulmonologist or attending physician.
Assess the impact of the device on the organisation of care. (2) | 3 years
  Duration of emergency, resuscitation, consultations and teleconsultations with the pulmonologist or attending physician.
Assess the impact of the device on the organisation of care. (3) | 3 years
  Number and nature of follow-up examinations and new pathologies detected during follow-up.
Assess the impact of the device on the quality of support. (1) | 3 years
  Number and nature of prescribed pharmacological treatments and prescribed oxygen therapy.
Assess the impact of the device on the quality of support. (3) | 3 years
  Duration of prescribed pharmacological treatments and prescribed oxygen therapy.
Assess patient and caregiver satisfaction with the device. (1) | 1 year
  Subjective assessment by the patient of the device, the reassurance provided by the device, the assistance to resume physical activity provided by the device, obtained using satisfaction questionnaires at M6 and M12.
Assess patient and caregiver satisfaction with the device. (2) | 1 year
  Subjective assessment by the patient of the overall quality of follow-up obtained using a detailed questionnaire (Likert scale) and an open-ended question about possible improvements at M6 and M12.
Assess patient and caregiver satisfaction with the device. (3) | 1 year
  Subjective assessment by caregivers of the Bora Care solution's impact on patient care using questions about organizational impacts and improved quality of care provided by the device, obtained using a satisfaction questionnaire at M6 and M12.
Evaluate the performance of the warning device in the early detection of exacerbations. | 3 years
  The number and nature of the alerts issued by the Bora Care solution, the number and nature of the actions taken following the alert specified in the alert management tool in the Bora Connect tool.
Identify new markers of exacerbations or other clinical events. | 3 years
  Alert performance in detecting exacerbations and other medical events by calculating alert sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ROCHE, MD, Principal Investigator — Hôpital Cochin, AP-HP
Locations (10):
- France (10):
  - CHU de Brest, Brest, Brittany Region
  - Centre Hospitalier Bretagne Atlantique, Vannes, Brittany Region
  - Centre Hospitalier de Chartres, Le Coudray, Centre-Val de Loire
  - Centre Hospitalier Verdun, Verdun, Grand Est
  - Groupement des Hôpitaux de l'Institut Catholique de Lille (GHICL), Lille, Hauts-de-France
  - Clinique du Millénaire, Montpellier, Occitanie
  - Centre Hospitalier Universitaire de Toulouse, Toulouse, Occitanie
  - Hôpital Européen Marseille, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hôpital de la Pitié Salpêtrière - AP-HP, Paris, Île-de-France Region
  - Hôpital Cochin - AP-HP, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No
Not applicable. Data are not intended to be shared with other researchers.